CLINICAL TRIAL: NCT00857714
Title: Lapatinib in the Treatment of Ductal Carcinoma in Situ of the Breast
Brief Title: Lapatinib for Treatment of Ductal Carcinoma In Situ (DCIS) of the Breast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Indiana University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0812-11
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Ductal Carcinoma in Situ
Keywords: DCIS; breast
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lapatinib — 1500 mg lapatinib for 14-21 days
  Other Names: Tykerb

SUMMARY:
The purpose of this study is to establish the utility of lapatinib in the treatment of DCIS, particularly ER-negative DCIS.

DETAILED DESCRIPTION:
Ductal carcinoma in situ (DCIS) of the breast is a pre-malignant lesion of the breast, which is associated with a marked increase in the likelihood of developing invasive breast cancer. Since DCIS tends to be associated with microcalcifications, it is detected with an increased frequency in patients being screened with mammographic techniques. The treatment of DCIS is based on a number of parameters; local treatment depends on the size of the lesion, grade and margins. The only systemic treatment currently available is in the form of endocrine therapy; it depends on the expression of estrogen receptor (ER). Randomized trials have shown that the treatment of DCIS with breast conserving therapy and radiation is as effective as simple mastectomy.

The efficacy of tamoxifen in reducing the incidence of further invasive or non-invasive breast cancer has been established. In addition to surgery (with or without radiation), patients with ER positive disease also receive anti-estrogen therapy. Current guidelines do not recommend any additional therapy for ER-negative DCIS.

The rationale for the proposed study is based on the observations that HER2 is expressed at high levels in higher grades of DCIS, which typically lack ER. In addition, an inverse relationship between ER expression and the expression of EGFR has also been demonstrated. Lapatinib is active against both these receptors and may have therapeutic action in ER negative DCIS.

We propose to treat the patients with drug in the interval between biopsy diagnosis and definitive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Patients with operable, biopsy-proven DCIS detected by screening mammography.
3. ER/PR negative DCIS.
4. DCIS that is positive for HER-2 &/or EGFR, which is defined as IHC 3+.
5. Women of childbearing potential willing to use an accepted and effective barrier method of contraception.
6. ECOG performance status ≤2
7. Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Patients must have normal organ and marrow function as defined below:

   * leukocytes ≥3,000/microL
   * absolute neutrophil count ≥1,500/microL
   * platelets ≥100,000/microL
   * total bilirubin within normal institutional limits
   * AST (SGOT)/ALT(SGPT) within normal institutional limits
   * creatinine within normal institutional limits OR creatinine clearance greater than or equal to 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal (using Cockcroft-Gault formula)

Exclusion Criteria:

1. Invasive breast cancer
2. ER+ or PR+ DCIS
3. Pregnant or breast feeding women
4. Patients who have had prior treatment with EGFR targeting therapies.
5. Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy. In addition, all herbal (alternative) medicines are excluded one week before starting lapatinib and for the duration of lapatinib therapy.
6. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
7. HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib.
8. Have ANY hepatic or biliary disease or dysfunction.
9. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
10. Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors.
11. ANY history of cardiac disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Badve, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty patients were expected for this trial but it stopped at one patient due to difficulty with recruitment.
Groups:
- 1500 mg Lapatinib for 14-21 Days: Patients took 1500 mg Lapatinib for 14-21 days until surgical excision.
Period: Overall Study
Arm/Group | 1500 mg Lapatinib for 14-21 Days
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1500 mg Lapatinib for 14-21 Days
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (NA) — Only one patient available; standard deviation cannot be calculated.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Where Gene Signature Was Obtained.
Description: Number of patients where gene signature was obtained. This was used to identify gene signature that denotes effect of lapatinib therapy in breast cancer cell lines and to assess effect of lapatinib therapy in patients with ductal carinoma in situ of the breast using the gene signature developed as a surrogate marker.
Time Frame: Up to 60 days
Measure: Number; unit: participants
Arm/Group | 1500 mg Lapatinib for 14-21 Days
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: Number of Patients With Toxicity Associated With Short Therapy With Lapatinib.
Description: Number of patients with toxicity associated with short therapy with lapatinib will be reported.
Time Frame: Up to 60 days
Measure: Number; unit: participants
Arm/Group | 1500 mg Lapatinib for 14-21 Days
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: Up to 60 days
Arm/Group | 1500 mg Lapatinib for 14-21 Days
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1500 mg Lapatinib for 14-21 Days (N=1)
Wound complication (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1500 mg Lapatinib for 14-21 Days (N=1)
skin rash (Skin and subcutaneous tissue disorders) | 1
nail changes (Skin and subcutaneous tissue disorders) | 1
mouth sores (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
cramping (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes